CLINICAL TRIAL: NCT01664091
Title: An Evaluation of Cosmetic Results and Toxicity in the Use of Post-Mastectomy Immediate Reconstruction With a Tissue Expander and Acellular Dermal Matrix Followed by Radiation Therapy
Brief Title: Cosmetic Result/Toxicity in Post-Mastectomy Immediate Reconstruction Expander+RT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Julia S. Wong, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-254
Record Dates: First submitted 2011-06-22; First posted 2012-08-14 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-08-26 (Actual); Status verified 2019-08

CONDITIONS: Breast Cancer
Keywords: tissue expander; acellular dermal matrix
MeSH Terms: conditions — Breast Neoplasms | interventions — Tissue Expansion Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TE-ADM with PMRT (Experimental): Participants received immediate breast reconstruction using a sub-muscular tissue expander (TE) and acellular dermal matrix (ADM) sling placed during the same surgery. This was followed by post-mastectomy radiation therapy (PMRT) no sooner than a minimum of 6 weeks and optimally 6 months, if adjuvant chemotherapy was required. The prescribed chest-wall dose was 50 -50.4 gray (Gy) in 25-28 fractions given once daily over 5-7 weeks with a 0.5-centimeter (cm) bolus to the scar every other day. Permanent reconstruction was performed at least 5 months after completion of PMRT.
  Interventions: Radiation: post-mastectomy radiation therapy (PMRT); Device: tissue expander (TE); Device: acellular dermal matrix (ADM)

INTERVENTIONS:
Radiation: post-mastectomy radiation therapy (PMRT)
Device: tissue expander (TE)
Device: acellular dermal matrix (ADM)

SUMMARY:
This research study is being done to carefully evaluate the effect of giving radiation therapy after temporary breast reconstruction. The investigators want to see if this type of reconstruction combined with radiation will look better (once the final reconstruction has been completed) and will reduce the risk that the participant will develop complications that sometimes occur with other kinds of reconstruction procedures. The investigators also want to know if it is easier to give the radiation with this type of reconstruction than with other kinds of reconstruction procedures. The reconstruction procedure involves the temporary use of a tissue expander and an acellular dermal matrix (ADM).

DETAILED DESCRIPTION:
* ADMs have been used in combination with a tissue expander and radiotherapy but have not been studied formally in terms of their ability to avoid complications sometimes seen with other methods of reconstruction and improve the delivery of the radiation. The only difference between being on the study and not being on the study is that the research team will analyze the records of those who participate to see how easy it was to give the radiation, how good the cosmetic outcome of the reconstruction is and what, if any, complications occured.
* A minimum of 6 weeks between the surgery and the start of radiation therapy is required to allow for adequate healing. Often this interval will be longer, as many patients will receive chemotherapy in the interim. There is no maximum time from surgery to radiation.
* Around the time of radiation planning, the radiation oncologist and plastic surgeon will agree upon how much deflation of the tissue expander will be required to permit simulation of the radiation therapy.
* Radiation therapy to the chest wall (with or without adjacent lymph nodes) will be given once daily Monday through Friday over 5-7 weeks.
* After the completion of the radiation therapy, the tissue expander will be re-expanded and eventually replaced by the permanent implant or flap reconstruction at the discretion of the plastic surgeon.
* Participants will be expected to return to the Radiation Oncology Clinic for follow-up visits 6, 12, 18 and 24 months after the end of the radiation therapy. Evaluation of cosmetic results and complications will be done at these visits using a recognized scoring system and photographs taken at each time point and scored for specific items (necrosis, telangiectasia, etc).

ELIGIBILITY:
Inclusion Criteria:

* Patients must have newly diagnosed, clinical Stage I-III breast cancer with T1-T3 invasive tumors recently treated with mastectomy
* Patients must have had immediate reconstruction with a TE and ADM
* Participants must be candidates for postmastectomy radiation therapy (RT). Postmastectomy RT routinely is indicated for patients with pathologically-staged T3N1 (or higher stage) tumors, T1-T2 tumors with 4 or more positive nodes, some T1-T2 tumors with 1-3 positive nodes, and, infrequently, for some N0 tumors
* Axillary nodes may be positive or negative
* Microscopically positive margins are permitted
* Systemic therapy as recommended by a medical oncologist, pre-or post-mastectomy, is permitted
* Patients must agree to return for scheduled follow-up visits with their radiation oncologist 6, 12, 18 and 24 months after RT (+/- 1 month)
* 18 years of age or older

Exclusion Criteria:

* Participants with T4 tumors
* Participants with recurrent breast cancer or a history of prior breast RT
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* Individuals with a history of a different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 5 years and are deemed by the investigator to be at low risk for recurrence of that malignancy. Individuals with the following cancers are eligible if diagnosed and treated within the past 5 years: cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin
* HIV-positive individuals on combination antiretroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julia Wong, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants enrolled from September 2009 through September 2012.
Groups:
- TE-ADM With PMRT: Participants received immediate breast reconstruction using a sub-muscular tissue expander (TE) and acellular dermal matrix (ADM) sling placed during the same surgery. This was followed by post-mastectomy radiation therapy (PMRT) no sooner than a minimum of 6 weeks and optimally 6 months, if adjuvant chemotherapy was required. The prescribed chest-wall dose was 50 -50.4 gray (Gy) in 25-28 fractions given once daily over 5-7 weeks with a 0.5-centimeter (cm) bolus to the scar every other day. Permanent reconstruction was performed at least 6 months after completion of PMRT.
Period: Overall Study
Arm/Group | TE-ADM With PMRT
Started | 32
Completed | 26
Not Completed | 6
Not completed — Death | 1
Not completed — Disease Progression | 2
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Groups:
- Tissue Expander and Acellular Dermal Matrix: immediate reconstruction with a TE and ADM followed by PMRT
  radiation: The prescribed chest-wall dose will be 50 - 50.4 Gy in 25-28 fractions, given once daily over 5-7 weeks.
Arm/Group | Tissue Expander and Acellular Dermal Matrix
Number analyzed (Participants) | 32
Age, Continuous [Median (Full Range); unit: years] | 42.3 [24.6 to 63.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Breast Cancer Laterality [Count of Participants; unit: Participants]
  Left | 15
  Right | 17
Mastectomy (unilateral, bilateral) [Count of Participants; unit: Participants]
  Unilateral | 18
  Bilateral | 14
Number of Lymph Nodes Excised [Median (Full Range); unit: lymph nodes] — Per Table 1 [Clinical and Treatment Characteristiscs], 'Lymph nodes' is a baseline variable further broken down to : 'No. Lymph Nodes involved' and 'No. Lymph Nodes excised'.
  For further information please reference Atkins et al. Effects of Postmastectomy Radiation Therapy on Immediate Tissue Expander and Acellular Dermal Matrix Reconstruction: Results of a Prospective Clinical Trial.
  lymph nodes | 11 [1 to 38]
Number of Lymph Nodes Involved [Median (Full Range); unit: lymph nodes] — Per Table 1 [Clinical and Treatment Characteristiscs], 'Lymph nodes' is a baseline variable further broken down to : 'No. Lymph Nodes involved' and 'No. Lymph Nodes excised'.
  For further information please reference Atkins et al. Effects of Postmastectomy Radiation Therapy on Immediate Tissue Expander and Acellular Dermal Matrix Reconstruction: Results of a Prospective Clinical Trial.
  lymph nodes | 2 [0 to 23]

OUTCOME MEASURES:

1. Primary Outcome: Success Rate
Description: Success rate was defined as the percentage of participants experiencing all of the following: 1) completion of PMRT and placement of the permanent implant and/or flap reconstruction; 2) no major complications (infection requiring hospitalization, major revisions, early/severe capsular contracture, or pain requiring implant removal); and 3) a physician-reported 'excellent' or 'good' cosmetic result (not 'fair' or 'poor') at 2 years following PMRT (requiring a stable reconstruction with good symmetry and contour relative to the contralateral breast).
Time Frame: 2 years
Population: The analysis population is comprised of the evaluable subset of participants with complete 2 year follow-up data.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | TE-ADM With PMRT
Number analyzed (Participants) | 26
percentage of participants | 65.4 [44.3 to 82.8]

2. Secondary Outcome: Lung Dose-Volume
Description: Lung dose-volumes were assessed as a percentage of the ipsilateral lung irradiated via dose-volume histograms.
Time Frame: Lung dose-volume was measured at the end of radiation therapy which was up to 11 weeks from enrollment in this study cohort.
Population: The analysis population is comprised of all enrolled participants.
Measure: Median (Full Range); unit: percentage radiation dose to lung
Arm/Group | TE-ADM With PMRT
Number analyzed (Participants) | 32
percentage radiation dose to lung | 28.7 [6.8 to 38.1]

3. Secondary Outcome: Cosmetic Score
Description: Cosmesis was measured by means of strict photographic analysis using five views (frontal, right and left lateral, and right and left quarter views) and independent assessment of the results by a plastic surgeon or radiation oncologist who has not treated the patient. Cosmetic score was defined in 4 categories: Excellent = treated breast looks essentially the same as the opposite breast; Good = minimal but identifiable result of treatment; Fair = significant effects of radiation therapy noted; Poor = severe normal tissue sequelae.
Time Frame: 2 years
Population: The analysis population is comprised of the evaluable subset of participants with complete 2 year follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | TE-ADM With PMRT
Number analyzed (Participants) | 24
Participants
  Excellent | 2
  Good | 17
  Fair | 5
  Poor | 0

4. Secondary Outcome: Baker Classification Peak Score
Description: An independent assessment of contracture was conducted by a plastic surgeon or radiation oncologist who had not treated the participant. Photographic analysis incorporated five views (frontal, right and left lateral, and right and left quarter views). Baker classification was used to score the extent of contracture: Class IA-absolutely natural, cannot tell breast was reconstructed; Class IB-soft, but the implant is detectable by physical examination or inspection because of mastectomy; Class II-mildly firm reconstructed breast with an implant that may be visible and detectable by physical examination; Class III-moderately firm reconstructed breast with readily detectable implant, but the result may still be acceptable; or Class IV-severe capsular contracture with an unacceptable aesthetic outcome and/or significant patient symptoms requiring surgical intervention.
Time Frame: Assessed up to 2 years post PMRT
Population: The analysis population excludes 1 participant lost-to follow-up who left the country immediately following PMRT.
Measure: Count of Participants; unit: Participants
Arm/Group | TE-ADM With PMRT
Number analyzed (Participants) | 31
Participants
  IA | 0
  IB | 1
  II | 15
  III | 14
  IV | 1

5. Secondary Outcome: Baker Classification 2-Year Score
Description: as for outcome 4
Time Frame: 2 Years
Population: The analysis population is comprised of the evaluable subset of participants with complete 2 year follow-up data.
Measure: Count of Participants; unit: Participants
Arm/Group | TE-ADM With PMRT
Number analyzed (Participants) | 22
Participants
  IA | 0
  IB | 8
  II | 7
  III | 7
  IV | 0

ADVERSE EVENTS:
Time Frame: Specific adverse events (AEs) as listed were evaluated and reported on the follow-up and cosmetic evaluation case report form at 6-, 12-, 18- and 24 months post RT. AEs were graded according to 5 classifications: mild, mild-moderate, moderate, moderate-severe and severe. Serious AEs were defined as AEs with a classification of moderate-severe or severe and other AEs with a classification of mild, mild-moderate or moderate.
Description: The analysis population excludes 1 participant lost-to follow-up who left the country immediately following PMRT.
Arm/Group | TE-ADM With PMRT
All-Cause Mortality (participants affected / at risk) | 1/31
Serious Adverse Events (participants affected / at risk) | 4/31
Other Adverse Events (participants affected / at risk) | 30/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TE-ADM With PMRT (N=31)
Delayed Healing Wound (Skin and subcutaneous tissue disorders) | 1
Infection (Infections and infestations) | 1
Deflation (Reproductive system and breast disorders) | 1
Asymmetry (Reproductive system and breast disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TE-ADM With PMRT (N=31)
Delayed Healing (Skin and subcutaneous tissue disorders) | 1
Skin Ischemia (Skin and subcutaneous tissue disorders) | 2
Infection (Infections and infestations) | 1
Chronic Drainage (Skin and subcutaneous tissue disorders) | 2
Pain/costochondritis (Musculoskeletal and connective tissue disorders) | 19
Asymmetry (Reproductive system and breast disorders) | 26
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 15
Deflation (Reproductive system and breast disorders) | 3

LIMITATIONS AND CAVEATS:
The major limitation of this study was its small sample size and its single arm nature.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No